CLINICAL TRIAL: NCT05522400
Title: Virtual Reality (VR) and Human Computer Interaction System in the Early Stage of ICU Patients Development and Application of Rehabilitation Exercise
Brief Title: Development and Application of Virtual Reality (VR) and Human Computer Interaction System in the ICU Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020ZSLC68
Record Dates: First submitted 2021-11-30; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Rehabilitation Exercise of ICU Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: Virtual Reality (VR) and human computer interaction system
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Virtual Reality (VR) and human computer interaction system — The experimental group used VR technology and human-computer interaction system for exercise, while the control group used traditional exercise program
  Arms: intervention group

SUMMARY:
By developing of VR and human computer interaction system of early rehabilitation exercise for ICU patients, this project aims to construct virtual scenes and realize the interaction between ICU patients and virtual scenes during active rehabilitation training for critically ill patients in long-term bed. This project can increase the patient's willingness to exercise rehabilitation, improve the training effect and improve clinical outcomes in critically ill patients.

ELIGIBILITY:
* Inclusion Criteria:

  * Over 18 years of age
  * Voluntary participation
* Exclusion Criteria:

  * Unable to walk independently before admission to ICU;
  * High dose of vasoactive drugs to maintain vital signs;
  * Acute stroke;
  * Upper limb fractures or amputations;
  * Patients with spinal fracture or pathological fracture;
  * Patients who have been hospitalized for 30 days or more before admission to ICU;
  * Plan to move out of ICU within 24 hours; In palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of the ICU-acquired asthenia | up to 2 weeks
  during ICU stay
Average daily physical activity time | up to 2 weeks
  during ICU stay
length of ICU stay | up to 2 weeks
  during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Wenyan PAN, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China